CLINICAL TRIAL: NCT04828733
Title: A Randomized Controlled Trial of Laparoscopic One Anastomosis Gastric Bypass With Excluded Stomach Fundoplication: FundoRingOAGB Versus NissenOAGB Versus OAGB Without Fundoplication for Treating Morbid Obesity and GERD
Brief Title: One Anastomosis Gastric Bypass With Excluded Stomach Fundoplication: FundoRing vs Nissen vs OAGB Without Fundoplication
Acronym: FundoRing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Society of Bariatric and Metabolic Surgeons of Kazakhstan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FundoRing vs Nissen
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Obesity; GERD
Keywords: Obesity; GERD; Gastric bypass; Fundoplication; Nissen; FundoRing
MeSH Terms: conditions — Obesity; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OAGB + SCP + FundoRing (Experimental): laparoscopic one anastomosis gastric bypass with excluded stomach fundoplication: FundoRingOAGB and suture cruroplasty
  Interventions: Procedure: laparoscopic one anastomosis gastric bypass with excluded stomach fundoplication: FundoRingOAGB and suture cruroplasty
- OAGB + SCP + NF (Active Comparator): laparoscopic one anastomosis gastric bypass with excluded stomach Nissen fundoplication and suture cruroplasty
  Interventions: Procedure: laparoscopic one anastomosis gastric bypass with excluded stomach Nissen fundoplication and suture cruroplasty
- OAGB + SCP (Active Comparator): laparoscopic one anastomosis gastric bypass without excluded stomach fundoplication and only suture cruroplasty
  Interventions: Procedure: Standard laparoscopic one anastomosis gastric bypass with cruroplasty. Not used fundoplication.

INTERVENTIONS:
Procedure: laparoscopic one anastomosis gastric bypass with excluded stomach fundoplication: FundoRingOAGB and suture cruroplasty — Laparoscopic gastric bypass with suture cruroplasty and excluded stomach fundoplication use FundoRing method.
  Arms: OAGB + SCP + FundoRing
Procedure: laparoscopic one anastomosis gastric bypass with excluded stomach Nissen fundoplication and suture cruroplasty — Laparoscopic gastric bypass with suture cruroplasty and excluded stomach fundoplication use the Nissen method.
  Arms: OAGB + SCP + NF
Procedure: Standard laparoscopic one anastomosis gastric bypass with cruroplasty. Not used fundoplication. — Laparoscopic gastric bypass with only suture cruroplasty without fundoplication
  Arms: OAGB + SCP

SUMMARY:
Background and study aims:

Currently, one anastomosis Gastric Bypass (OAGB) is a common bariatric procedure.

Obesity and gastroesophageal reflux disease (GERD) are steadily increasing world weight and antireflux surgery must be performed simultaneously with bariatric surgery in obese patients. In these cases, most often for GERD patients OAGB procedures only with hiatus cruroraphy is performed.

The goal of this randomized controlled clinical trial is to compare bariatric and antireflux results after OAGB plus suture cruroplasty with FundoRing (n=50) versus Nissen fundoplication (n=50) and versus without total fundoplication (n=50) for patients with morbid obesity and GERD.

The main questions it aims to answer are:

* What is the impact of wrapping the fundus of the excluded part of the stomach use FundoRing method in the experimental group against developing reflux esophagitis compare impact standard Nissen in OAGB?
* What is the impact of excluded stomach fundoplication on weight loss in FundoRing group versus standard Nissen group in OAGB?

Methods: Adult participants (n=150) are randomly allocated to one of three groups:

Experimental surgical bariatric procedure in the first (A) group: patients (n=50) undergo the laparoscopic one anastomosis gastric bypass with excluded stomach fundoplication: FundoRingOAGB and suture cruroplasty (OAGB + SCP + FundoRing); Active comparator surgical bariatric procedure in the second (B) group: patients (n=50) undergo the laparoscopic one anastomosis gastric bypass with excluded stomach Nissen fundoplication and suture cruroplasty (OAGB + SCP +NF).

Active comparator surgical bariatric procedure in the second (C) group: patients (n=50) undergo laparoscopic one anastomosis gastric bypass without excluded stomach fundoplication and only suture cruroplasty (OAGB + SCP). All patients are then followed up 12, 24, and 36 months after surgery where the changing body mass index and change of GERD symptoms (GERD-HRQL).

DETAILED DESCRIPTION:
One anastomosis Gastric Bypass/Mini Gastric Bypass (OAGB/MGB) is gaining popularity as a primary surgical treatment for morbid obesity. The total fundoplication is the gold standard for treating GERD. Morbid obesity and GERD require simultaneous surgical treatment.

The aim study is to compare bariatric and antireflux results after OAGB/MGB plus suture cruroplasty (SCP) with FundoRing versus Nissen fundoplication and versus without total fundoplication.

Adult participants (n=150) are randomly allocated to one of three groups:

Experimental surgical bariatric procedure in the first (A) group: patients (n=50) undergo the laparoscopic one anastomosis gastric bypass with excluded stomach fundoplication: FundoRingOAGB and suture cruroplasty (OAGB + SCP + FundoRing); Active comparator surgical bariatric procedure in the second (B) group: patients (n=50) undergo the laparoscopic one anastomosis gastric bypass with excluded stomach Nissen fundoplication and suture cruroplasty (OAGB + SCP +NF).

Active comparator surgical bariatric procedure in the second (C) group: patients (n=50) undergo laparoscopic one anastomosis gastric bypass without excluded stomach fundoplication and only suture cruroplasty (OAGB + SCP). All patients are then followed up 12, 24, 36 months after surgery where record the changing body mass index and change of GERD symptoms (GERD-HRQL).

ELIGIBILITY:
Inclusion Criteria:

* Class I- III obesity (BMI 30.0-50.0 kg/m)
* Patients with GERD A or B grade of reflux esophagitis (LA grade) after treatment PPI
* Hiatal hernia (HH) <5 cm
* ASA grading 1-2
* Age 18-60 years old.

Exclusion Criteria:

* Giant hiatal hernia (HH) >5 cm
* Esophageal shortening
* Patients with C or D grade of RE (reflux esophagitis)
* Previously surgery on the stomach or esophagus
* Psychiatric illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Change of body mass index | Baseline, at 12, 24, 36 months after surgery
  The measure is assessing a change of body mass index. Weight (kg) and height (cm) will be combined with the report of measurement by body mass index (BMI) kg/m2.
Change of GERD symptoms (GERD-HRQL) | 12, 24, 36 months after surgery
  Success; ≥50% improvement in the baseline GERD-HRQL score Failure; <50% improvement in the baseline GERD-HRQL score at 12,24, 36 months.

CONTACTS AND LOCATIONS:
Overall Officials: Oral Ospanov, Professor, Principal Investigator — President of Society of Bariatric and Metabolic Surgeons of Kazakhstan" (SBMSK)
Locations (1):
- Oral Ospanov, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ospanov O, Zharov N, Yelembayev B, Duysenov G, Volchkova I, Sultanov K, Mustafin A. A Three-Arm Randomized Controlled Trial of Primary One-Anastomosis Gastric Bypass: With FundoRing or Nissen Fundoplications vs. without Fundoplication for the Treatment of Obesity and Gastroesophageal Reflux Disease. Medicina (Kaunas). 2024 Feb 27;60(3):405. doi: 10.3390/medicina60030405. PMID 38541131